CLINICAL TRIAL: NCT05575531
Title: The Effect of Modified Early Warning Scoring System and Nursing Guide Practices on Postoperative Patient Outcomes
Brief Title: Evaluation of the Modified Early Warning Scoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, SELDA MERT, Assist. Prof. Dr., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAEK/17.bI.02
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-03

CONDITIONS: Clinical Deterioration; Postoperative Complications; Nurse's Role
Keywords: Clinical deterioration; early warning score; nursing assessment; postoperative care; surgical nursing
MeSH Terms: conditions — Clinical Deterioration; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomized-controlled clinical trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): MEWSS and Nursing Guide Application will be used in the study group. MEWSS: The Modified Early Warning Score (MEWS) consists of a simple to use algorithm based on physiological parameters such as heart rate, respiratory rate, systolic blood pressure, temperature and level of consciousness.
  Nursing Guide Application (NGA): According to the follow-up carried out in this study: If the patient's MEWSS is 4 or below, a ten-minute follow-up was performed. If the MEWSS is five, then five-minute follow-up is passed, and if the score has not changed as a result of the follow-ups, five-minute follow-ups are continued. If the score decreased to four or less, ten-minute follow-up was started, if the score increased, five-minute follow-ups were continued, and the emergency team was informed and the patient was evaluated (the emergency team was informed about the study).
  Interventions: Other: MEWSS and Nursing Guide Application
- Control Group (No Intervention): In the control group, the patients followed according to the Modified Early Warning Scoring System received routine care in the clinic.

INTERVENTIONS:
Other: MEWSS and Nursing Guide Application — MEWSS and Nursing Guide application will be used for the patients in the experimental group. According to the Nursing Guide application, patients with MEWS above 4 will be monitored every 5 minutes, while those with a score below 4 will be monitored for 10 minutes. will be followed intermittently. Nursing interventions will be made in accordance with the problems experienced by patients with a score above 4.
  Arms: Experimental Group

SUMMARY:
In this study, it was aimed to determine the effect of HRU and HG on patient outcomes in the care process in surgical patients followed according to MEUSS.

The sample of the study, which was conducted as a randomized-controlled clinical trial, consisted of 252 patients who underwent surgical intervention under general anesthesia in a university hospital between 29 July 2022 and 31 October 2022.

DETAILED DESCRIPTION:
Postoperative patients are at risk of clinical worsening and minimizing this is vital. Nurses play a vital role in the early detection and management of clinical deterioration as they are the group of professionals with the highest patient contact. MEUSS is stated as a simple risk management tool based on physiological parameters that can allow early detection of clinical deterioration and initiation of the relevant intervention, improving the quality of care and patient safety provided to surgical patients.

In this study, with a larger sample, patients will be followed up with MEUSS and a nursing guide for 2 hours in the clinic where they are transferred both after and after ASBU. Our study is a research with the highest sample in this field, in which patients are followed for the longest period of time, and it is thought that MEUSS and nursing guide applications can identify risky patients in the postoperative period and reduce postoperative complications with strict follow-up applied to these patients. The aim of this study; To determine the effect of Nursing Guide Practice (HRU) and Nursing Interventions (HG) on patient outcomes in the care process in surgical patients followed according to MEUSS.

ELIGIBILITY:
Inclusion Criteria:

* Having operated under general anesthesia
* transferred to the post-anesthesia care unit (ASBU) and then to the service/ICU followed for 2 hours,
* between 18-65 years old,
* who have not had an operation with general anesthesia in the last six months,
* no serious life-threatening complications developed during surgery,
* patients willing to participate in the study

Exclusion Criteria:

* data unavailable,
* complications during surgery,
* patients who did not undergo general anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Effects of MEWSS and NGA use on complications and clinical status | From the first 5 minutes when the patient comes to the post-anesthesia care unit to the end of the second hour
  Length of stay in ASBU (minutes), complications developed in ASBU, intervention time to complications (minutes), and where it was transferred after ASBU (clinical or intensive care unit)
Effect of MEWSS and NGA use on vital signs and MEWS | From the first 5 minutes when the patient comes to the post-anesthesia care unit to the end of the second hour
  Heart rate (beats per minute), respiratory rate (respiratory rate / min.), systolic blood pressure (mmHg), temperature (centigrade degree -°C), level of consciousness (AVPU) and the score obtained from these measurements show MEWS.
Effect of MEWSS and NGA use on nursing interventions | From the first 5 minutes when the patient comes to the post-anesthesia care unit to the end of the second hour
  Nursing interventions include practices such as oxygen saturation, blood pressure, pulse, respiration, body temperature, alertness, pain monitoring by nurses, positioning and giving medication.

CONTACTS AND LOCATIONS:
Overall Officials: Selda MERT, Assist.Dr., Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)